CLINICAL TRIAL: NCT05335837
Title: Postoperative Recovery Time in Inguinal Hernia Repair Under Ilioinguinal, Iliohypogastric Nerve Block and Sedation Versus General Anesthesia: a Propensity Score Matched-cohort Retrospective Study
Brief Title: Ilioinguinal/Iliohypogastric Block for Inguinal Hernia Repair
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Cheng Lin, Clinical Professor, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Other Study IDs: 119564
Record Dates: First submitted 2022-04-09; First posted 2022-04-19 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Anesthesia
MeSH Terms: interventions — Anesthesia, Conduction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- General Anesthesia: patients received general anesthesia for inguinal hernia repair
- Regional Anesthesia and Sedation: patients received ilioinguinal/iliohypogastric nerve blocks and sedation for inguinal hernia repair
  Interventions: Procedure: Regional Anesthesia and Sedation

INTERVENTIONS:
Procedure: Regional Anesthesia and Sedation — Preoperative ilioinguinal/iliohypogastric nerve block and moderate to deep intraoperative sedation.
  Groups: Regional Anesthesia and Sedation

SUMMARY:
Inguinal hernia have traditionally been done under general anesthesia. While safe, general anesthesia is associated with potential postoperative nausea/vomiting and drowsiness. Additionally, the recent COVID19 pandemic has heightened the precaution to avoid aerosol generating procedures (AGP) if possible. General anesthesia requires airway manipulation, thus necessitate performing an AGP. Recently, we began using peripheral nerve block and sedation as primary anesthetic technique for inguinal hernia repairs. While surgeon administered local anesthetic, also known as local infiltration, has been done for inguinal hernia repair, using specific nerve blocks and sedation has not been compared with general anesthesia. We believe the advantage of this novel technique can improve postoperative recovery. This retrospective study will compare the total hospital length of stay of those receiving nerve blocks and sedation as primary anesthetic techniques versus those with general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* American Society of Anesthesiologists (ASA) Physical Status I to III
* Body Mass Index (BMI) less than 45
* Single hernia repair, elective, ambulatory surgery

Exclusion Criteria:

* Opioid dependence (30 mg oral morphine equivalents daily or more)
* History of malignant hyperthermia
* Pregnancy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative recovery time | Time from exiting operating room to time ready for hospital discharge, up to 100 hours
  Time from exiting operating room to time ready for hospital discharge

SECONDARY OUTCOMES:
Preoperative time | Time from patient registration to entering operating room, up to 100 hours
  Time from patient registration to entering operating room
Intraoperative time | Time from entering to exiting operating room, up to 100 hours
  Time from entering to exiting operating room
Hospital length of stay | Time from patient registration to ready for hospital discharge, up to 100 hours
  Time from patient registration to ready for hospital discharge
Postoperative nausea vomiting | Time from exiting operating room to time ready for hospital discharge, up to 100 hours
  Associated symptoms of nausea vomiting, or received non-prophylactic antiemetics
Severe pain | Time from exiting operating room to time ready for hospital discharge, up to 100 hours
  Any incidence when patient rated pain at least 7 out of 10 numeric rating scale
Desaturation | Time from exiting operating room to time ready for hospital discharge, up to 100 hours
  Oxygen saturation below 90% with or without oxygen
Postoperative opioid dose | Time from exiting operating room to time ready for hospital discharge, up to 100 hours
  total postoperative opioid dose in oral morphine equivalents

CONTACTS AND LOCATIONS:
Locations (1):
- Cheng Lin, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided